CLINICAL TRIAL: NCT02962804
Title: Combination Radiation and PD-1 Inhibition in Metastatic or Recurrent RCC
Brief Title: Combination Radiation and PD-1 Inhibition in Metastatic or Recurrent Renal Cell Carcinoma (RCC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to competing trials. Stopped before IRB approval.
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016XSGURadPlusPD1RenalCC
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: kidney; renal cell; cancer; metastatic; recurrent
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Nivolumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab plus radiation (Experimental): Nivolumab plus radiation
  Interventions: Drug: Nivolumab; Radiation: Radiation

INTERVENTIONS:
Drug: Nivolumab — 240 mg per IV infusion over 60 minutes every 14 days (+/- 2 days) until disease progression or participant withdrawal from study
  Other Names: OPDIVO
Radiation: Radiation — Radiation to at least 1 site (up to 3) of primary or metastasis, 5 fractions - delivered over 2 weeks, starting 1-3 days post-nivolumab administration. Recommended dose range is 6 Gy-12 Gy per fraction.

SUMMARY:
There are two primary aims in the study: 1) to determine the tolerability and feasibility of combination hypofractionated radiation therapy and PD-1 inhibition with nivolumab, and 2) to determine the ability of hypofractionated radiation therapy to enhance response rate from PD-1 inhibition versus PD-1 inhibition alone by comparing the observed response rate under the combination therapy with a previously reported response rate under inhibition alone.

DETAILED DESCRIPTION:
Patients with metastatic or recurrent renal cell cancer who have progressed on standard Tyrosine Kinase Inhibitor (TKI) therapy and who have metastatic or primary tumors suitable for palliative radiation will be eligible for this study. Treatment will consist of nivolumab plus hypofractionated radiation therapy. The primary endpoint will be objective response rate, which will be compared against the historical control of 25% using nivolumab alone as established in the CHECKMATE 025 clinical trial. Patients will continue on nivolumab until disease progression or withdrawal of consent. Follow-up will continue for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed history of renal cell carcinoma (all variants are acceptable)
2. Progression or recurrence after at least one prior tyrosine kinase inhibitor therapy including, but not limited to: sunitinib, pazopanib, axitinib.
3. At least 1 site (primary or metastasis) amenable to hypofractionated radiation therapy and appropriate for radiation therapy as part of standard of care per medical, urologic or radiation oncologist discretion. NOTE: CT / MRI imaging to have been completed no more than 30 days before enrollment on study.

   Potential indications for radiation therapy include (but are not limited to):
   * Painful bone or soft tissue metastasis
   * Symptoms from mass effect caused by tumor
   * Prevention of impending symptoms from tumor
   * Hemoptysis due to tumor
   * Limited oligometastasis
   * Isolated region of progression
4. Patients with prior IL-2 treatment are eligible
5. At least 14 days since any prior therapy
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 3
7. Adequate organ and marrow function as defined below:

   * leukocytes ≥ 2,000/mcL
   * absolute neutrophil count ≥ 1,000/mcL
   * platelets ≥ 100,000/mcL
   * total bilirubin within normal institutional limits
   * AST(SGOT) ≤ 2.5 X institutional upper limit of normal
   * ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
8. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception. Men of child-bearing potential must not donate sperm while on this study and for 90 days after their last study treatment.

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Men who are trying to father a child.
3. Presence of a condition or abnormality that in the opinion of the study-delegated investigator would compromise the safety of the patient or the quality of the data.
4. Requirement for high dose steroids: dexamethasone > 2 mg per day or equivalent

   * NOTE: Per OPDIVO (Nivolumab) package insert, no formal pharmacokinetic drug-drug interaction studies have been conducted with OPDIVO (Nivolumab) - therefore, no other concomitant medications will exclude potential participants.
5. Life expectancy < 6 months.
6. Other active malignancy (patients with no evidence of disease (NED) or are in remission are eligible).
7. Patient has untreated brain metastases. Patients are eligible after documented stable or improved brain metastases at least 1 month after treatment of brain metastases.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to PD-1 Inhibitors used in study.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patients with active, known or suspected autoimmune disease (not including type 1 diabetes mellitus, hypothyroidism, skin disorders not requiring systemic treatment or conditions not expected to recur).
11. Patients with interstitial lung disease
12. Patients receiving concurrent other cancer-directed therapy including, but not limited to, Tyrosine Kinase Inhibitor (TKI), Mammalian Target Of Rapamycin (mTOR) inhibition and/or chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Every 3 months up to 2 years or progression
  Objective response rate (ORR) defined as the sum of partial response (PR) and complete response (CR). Timeframe will be best response from registration to end of treatment.

SECONDARY OUTCOMES:
ORR at irradiated sites | Every 3 months up to 2 years or progression
ORR at un-irradiated sites | Every 3 months up to 2 years or progression
Progression free survival (PFS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xinglei Shen, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States